CLINICAL TRIAL: NCT05033743
Title: Suppressive Antibacterial Therapy With Once-Weekly Secnidazole Granules to Prevent Recurrent Bacterial Vaginosis; A Pilot Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Lupin Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Chemen M. Neal, Assistant Clinical Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10283
Record Dates: First submitted 2021-08-09; First posted 2021-09-05 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Recurrent Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Secnidazole treatment
  Interventions: Drug: Secnidazole 2 GM Oral Granules

INTERVENTIONS:
Drug: Secnidazole 2 GM Oral Granules — Once weekly 2g oral secnidazole for 18 weeks

SUMMARY:
The purpose of this study is to test the effectiveness Secnidazole to treat recurrent BV. Secnidazole is approved for one-time use in acute BV. In this study, the drug will be used for recurrent BV, and given weekly for 18 weeks.

DETAILED DESCRIPTION:
A single-center prospective pilot study with once-weekly oral secnidazole granule treatment of acute condition for two-weeks followed by prophylactic treatment of asymptomatic responders with once-weekly secnidazole for 16 weeks, followed by no therapy for 12 weeks. The final follow-up evaluation is at week 28.

Eligible women with a current symptomatic bacterial vaginosis infection (> or = 3 Amsel criteria) and a history of at least 2 previous episodes of bacterial vaginosis in the past year will be enrolled in the open-label treatment study. All women will be treated with 2g of secnidazole granules orally once-weekly for 2 weeks. At the second visit, 3-5 days after completion of treatment, women who have a resolution of bacterial vaginosis (asymptomatic and < or = 2 Amsel criteria) will continue on once-weekly secnidazole for 16 weeks.

Patients will be evaluated every 4 weeks for recurrence of bacterial vaginosis. This will include questions about symptoms as well as a pelvic examination for assessment of vaginal discharge (> or = 3 Amsel criteria). We will also collect any information on other clinical evaluations for recurrence and the dates of diagnoses and types of treatments they may have received. Those who remain without recurrence during the 16-week suppressive phase will be followed for an additional 12 weeks off therapy, with assessment for recurrence at weeks 22 and 30. Throughout the study, data will be collected on participants' compliance and on the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Ability to consent in English
* Current symptomatic bacterial vaginosis infection
* History of at least 2 previous episodes of bacterial vaginosis in the past year

Exclusion Criteria:

* Current gynecologic infection or condition, including candida vaginitis, gonorrhea, chlamydia, trichomonas, desquamative inflammatory vaginitis, atrophic vaginitis.
* Pre-existing heart conditions
* Pre-existing neurological conditions
* Currently Pregnant or breastfeeding
* Women taking anticoagulants, lithium, metoclopramide, or disulfiram therapy
* Hypersensitivity to secnidazole or other drugs in the same class.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chemen Neal, MD, Principal Investigator — Assistant Professor
Locations (1):
- Indiana University Hospital - Coleman Center for Women, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 24
Completed | 20
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: prescribed once-weekly secnidazole for 16 weeks as prophylactic treatment
Groups:
- Secnidazole: prescribed once-weekly secnidazole for 16 weeks as prophylactic treatment
Arm/Group | Secnidazole
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 16
  Hispanic | 1
  White | 7
Region of Enrollment [Number; unit: participants]
  United States | 24
Bacterial Vaginosis (BV) episodes in prior 12 months [Mean (Standard Deviation); unit: episodes] — Population: 4 participants were withdrawn or lost to followup before this baseline measure was collected. These participants were excluded from analysis.
  episodes
    number analyzed (Participants) | 20
    (all) | 8.1 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Episode of Bacterial Vaginosis
Description: Overall failure rate as measured by the number of subjects with at least one episode of bacterial vaginosis in the 30 week follow-up period.
Time Frame: 30 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
Participants | 8

2. Primary Outcome: Probability of Failure at 210 Days
Description: To assess the efficacy of secnidazole, we estimated failure rates and 95% exact confidence intervals for initial treatment, suppression therapy following initial resolution of BV symptoms, and overall. For the time-to-failure analysis, time was defined as the number of days since the second visit where clinical resolution of initial BV was confirmed. The non-parametric maximum likelihood estimate (NPMLE) of the survival curve was estimated using the interval package in R to account for the interval censored data. Results are presented using an Amsel criteria score of as well as for BV diagnosis. All analyses were conducted using R 4.2.2 (R Core Team, 2020) in RStudio (RStudio Team 2021).
Time Frame: 210 days (30 weeks)
Population: The calculation only includes participants who began the suppression portion of the study and participants who were not withdrawn or lost to follow-up.
Measure: Number; unit: Probability
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Probability | 0.7051

3. Primary Outcome: The Number of Subjects That Failed Treatment in the Supressive Phase
Description: The probability of recurrence or treatment failure was calculated as time from the second visit in days. This timeframe is the suppressive therapy phase and was 30 weeks long.
Time Frame: 30 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 3

4. Secondary Outcome: Number of Subjects Who Experienced Recurrence 3-5 Days After Initial Treatment (Initial Treatment Was 2 Weeks Long)
Description: Recurrence was measured using the Amsel criteria. The Amsel criteria are: 1) Homogenous white discharge, 2) pH > 4.5, 3) amine odor (whiff) test, 4) clue cells on microscopy
Time Frame: 3-5 days after initial treatment after initial treatment of 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 20
Participants | 5

5. Secondary Outcome: Number of Subjects Who Experienced Recurrence 6 Weeks After Start of Initial Treatment
Description: as for outcome 4
Time Frame: week 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 0

6. Secondary Outcome: Number of Subjects Who Experienced Recurrence 10 Weeks After Start of Initial Treatment
Description: as for outcome 4
Time Frame: week 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 0

7. Secondary Outcome: Number of Subjects Who Experienced Recurrence 14 Weeks After Start of Initial Treatment
Description: as for outcome 4
Time Frame: week 14
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 1

8. Secondary Outcome: Number of Subjects Who Experienced Recurrence 18 Weeks After Start of Initial Treatment
Description: as for outcome 4
Time Frame: week 18
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 1

9. Secondary Outcome: Number of Subjects Who Experienced Recurrence 22 Weeks After Start of Initial Treatment
Description: as for outcome 4
Time Frame: week 22
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 2

10. Secondary Outcome: Number of Subjects Who Experienced Recurrence 30 Weeks After Start of Initial Treatment
Description: as for outcome 4
Time Frame: week 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 3

11. Other Pre Specified Outcome: Number of Participant With Compliance
Description: Subject compliance with the study medication, based on questionnaire that asked if the participant took the medication as scheduled and asked about side effects.
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 15

12. Other Pre Specified Outcome: Number of Participants With Tolerance
Description: Subject tolerance with the study medication, based on questionnaire that asked if the participant took the medication as scheduled and asked about side effects.
Time Frame: 18 weeks
Population: This number of participants includes all subjects, including lost to follow up and withdraws. Only one subject reported intolerance of the medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
Participants | 24

13. Other Pre Specified Outcome: Number of Adverse Events
Description: Number of adverse events that participants experienced
Time Frame: 30 weeks
Population: Analysis only includes participants who experienced an AE.
Measure: Number; unit: adverse events
Arm/Group | Treatment Group
Number analyzed (Participants) | 10
adverse events | 41

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=24)
Yeast Infection (Skin and subcutaneous tissue disorders) | 7 (12)
Headache (Nervous system disorders) | 2 (4)
Loose Stool (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (2)
UTI (Renal and urinary disorders) | 2 (2)
left lower quadrent pain (Gastrointestinal disorders) | 1 (1)
spotting (Reproductive system and breast disorders) | 1 (1)
urinary odor (Renal and urinary disorders) | 1 (1)
change in discharge (Reproductive system and breast disorders) | 1 (1)
COVID-19 infection (Infections and infestations) | 1 (1)
Post Operative Pulmonary Embolism (Vascular disorders) | 1 (1) — One patient suffered a pulmonary embolus while taking oral contraceptives and was in the immediate postoperative state. This was deemed unrelated to the study drug. She did not continue participation in the study due to anticoagulant use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT05033743/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT05033743/SAP_001.pdf
  • Informed Consent Form (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT05033743/ICF_002.pdf